CLINICAL TRIAL: NCT02918032
Title: International Registry Study of Neutral Lipid Storage Disease (NLSD) / Triglyceride Deposit Cardiomyovasculopathy (TGCV) and Related Diseases
Status: Recruiting | Type: Observational
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Responsible Party: Sponsor
Other Study IDs: TRICVD1315
Record Dates: First submitted 2016-08-04; First posted 2016-09-28 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Neutral Lipid Storage Disease
Keywords: Jordans anomaly; neutral lipid storage disease; triglyceride deposit cardiovasculopathy; ATGL gene; CGI-58 gene; primary triglyceride deposit cardiomyovasculopathy (TGCV); neutral lipid storage disease with myopathy (NLSD-M)
MeSH Terms: conditions — Chanarin-Dorfman Syndrome; Neutral Lipid Storage Disease with Myopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NLSD / TGCV: Patients who are diagnosed with NLSD / TGCV

SUMMARY:
This study aims to understand the state of onset of NLSD(neutral lipid storage disease) / TGCV(triglyceride deposit cardiovasculopathy) worldwide, background information of affected patients, and natural history of the disease, as well as exploring the prognostic factors and assessing the efficacy of disease-specific treatment.

DETAILED DESCRIPTION:
Since NLSD is a rare disease, its clinical manifestation and clinical course have not been sufficiently clarified. Also, the number of patients in each country is limited. As such, it is considered difficult to fully investigate this disease without international collaboration. Therefore, we have established the International Registry of NLSD / TGCV. Also, all patients with Jordans' anomaly of peripheral polymorphonuclear leukocytes are established as the subjects of entry when starting the registry, to allow entry of patients with NLSD due to genes other than mutations of ATGL and CGI-58 genes.

Time Perspective:This study is both Prospective (registering patients who are diagnosed with NLSD / TGCV) and Retrospective (registering only the medical record of previous patients).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with NLSD / TGCV

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are diagnosed with NLSD /TGCV (including adults only)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2014-01; Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Period from the diagnosis of NLSD / TGCV to death from any cause | 5 years
  This is the period from the date of diagnosis of NLSD / TGCV to the date of death from any cause. The last date of confirmation of survival will be used as the cut-off date for living patients and patients who are lost to follow-up.

SECONDARY OUTCOMES:
Serum CK(Creatine Kinase) level | 5 years
  Evaluating the serum CK level by measuring
Serum BNP(B-type Natriuretic Peptide) level | 5 years
  Evaluating serum BNP level by measuring
Serum AST(Aspartate transaminase) level | 5 years
  Evaluating serum AST level by measuring
Serum ALT(Alanine transaminase) level | 5 years
  Evaluating serum ALT level by measuring
Serum TG level | 5 years
  Evaluating serum TG level by measuring
Plasma glucose level | 5 years
  Evaluating plasma glucose level by measuring
HbA1c | 5 years
  Evaluating HbA1c by measuring
TSH(thyroid-stimulating hormone) | 5 years
  Evaluating TSH by measuring
Free T4 | 5 years
  Evaluating Free T4 by measuring
Ichthyosis | 5 years
  Presence / Absence of Ichthyosis within 5 years
Jordans' anomaly | 5 years
  Presence / Absence of Jordans' anomaly within 5 years
Neurosensory disorders | 5 years
  Presence / Absence of neurosensory disorders
Mental retardation | 5 years
  Presence / Absence of mental retardation
Hearing loss | 5 years
  Presence / Absence of hearing loss
Skeletal muscle (Musculoskeletal symptoms) | 5 years
  Presence / Absence of musculoskeletal symptoms
Skeletal muscle (Muscle weakness) | 5 years
  Presence / Absence of muscle weakness
Barthel Index | 5 years
  Evaluating activities of daily living by Barthel Index
Clinical findings of Heart | 5 years
  Presence / Absence of cardiac symptoms
Clinical findings of Liver | 5 years
  Presence / Absence of hepatomegaly
Clinical findings of Pancreas | 5 years
  Presence / Absence of diabetes mellitus
Manual muscle test | 5 years
  Evaluating muscles by Manual muscle test
Muscle biopsy | 5 years
  To evaluate lipid involvement and deposition
Myocardial biopsy | 5 years
  To evaluate lipid involvement and deposition
Skin biopsy | 5 years
  To evaluate lipid involvement and deposition
Respiratory function test | 5 years
  Evaluating muscles by Respiratory function test
6-minute walk distance | 5 years
  Evaluating heart function by 6-minute ｗalk distance
Treadmill endurance time | 5 years
  Evaluating heart function by treadmill endurance time
Cardiopulmonary exercise test | 5 years
  Evaluating heart function by cardiopulmonary exercise test
Skeletal muscle(CT) | 5 years
  Evaluating skeletal muscle using CT
Skeletal muscle(MRI) | 5 years
  Evaluating skeletal muscle using MRI
Skeletal muscle(electromyogram) | 5 years
  Evaluating skeletal muscle using electromyogram
Fatty liver(ultrasonography) | 5 years
  Evaluating fatty liver by ultrasonography
Thyroid(ultrasonography) | 5 years
  Evaluating thyroid by ultrasonography
Echocardiogram | 5 years
  Measuring echocardiogram
Cardiac CT | 5 years
  Measuring cardiac CT
Cardiac MRI | 5 years
  Measuring cardiac MRI
Coronary angiography | 5 years
  Measuring coronary angiography
Electrocardiogram | 5 years
  Measuring electrocardiogram
Holter monitoring | 5 years
  Measuring holter monitoring
BMIPP scintigram | 5 years
  Evaluating myocardial lipolysis

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Hirano, MD, Ph.D, Principal Investigator — Department of Cardiovascular Medicine, Faculty of Internal Medicine, Graduate School of Osaka University
Locations (15):
- United States (2):
  - Stanford University, Stanford, California
  - Columbia University, New York, New York
- University of Graz, Graz, Styria, Austria
- Peking University First Hospital, Beijing, Beijing Municipality, China
- Pitié-Salpêtrière Hospital, Paris, Paris, France
- Ludwig-Maximilians University, Munich, Bavaria, Germany
- Italy (4):
  - Sapienza University of Rome, Rome, Lazio
  - A.C.O. San Filippo Neri Hospital, Rome, Lazio
  - Catholic University, Milan, Lombardy
  - University of Padova, Padua, Veneto
- Japan (2):
  - Graduate School of Osaka University, Suita, Osaka
  - National Center of Neurology and Psychiatry, Kodaira, Tokyo
- Maastricht University, Maastricht, Limburg, Netherlands
- United Kingdom (2):
  - Harefield Hospital, Harefield, London
  - New Castle University, Newcastle upon Tyne, Tyne and Wear